CLINICAL TRIAL: NCT07359131
Title: Postoperative Assessment in TMJ Surgery: A Comparison of the Efficacy of Intraoperative Platelet-Rich Plasma and Platelet-Rich Fibrin Injections
Brief Title: Postoperative Assessment of Platelet-Rich Plasma and Platelet-Rich Fibrin in Temporomandibular Joint Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Jingping Wang, MD, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Jingping Wang, MD, Ph.D., Associate Professor Staff Anesthesiologist & Pain Physician, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Other Study IDs: 2024P003298
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 - Platelet-Rich Plasma injection therapy group: Patients who received Platelet-Rich Plasma injections during surgery.
- Group 2 - Platelet-Rich Fibrin injection therapy group: Patients who are receiving Platelet-Rich Fibrin injections during surgery.
- Group 3 - non injection therapy group: Patients who are not receiving Platelet-Rich Plasma nor Platelet-Rich Fibrin injections during surgery.

SUMMARY:
The goal of this observational study is to evaluate postoperative outcomes following temporomandibular joint (TMJ) surgery and to compare the effectiveness of intraoperative platelet-rich plasma (PRP) and platelet-rich fibrin (PRF) injections in patients with temporomandibular joint disorders.

The study includes adult patients who underwent TMJ surgery and received either PRP or PRF intraoperatively. The main questions this study aims to answer are:

Whether intraoperative PRP or PRF injection is associated with differences in postoperative pain intensity and recovery.

Whether PRP and PRF differ in their effects on postoperative jaw function, including maximum mouth opening and joint symptoms.

If there is a comparison group: Researchers will compare patients who received intraoperative PRP with those who received intraoperative PRF to assess differences in postoperative pain, functional outcomes, and joint-related symptoms.

Participants will:

Have their existing medical records reviewed retrospectively.

Provide postoperative outcome data derived from routine clinical follow-up, with no prospective recruitment or intervention.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 to 75 years (inclusive)

Underwent unilateral or bilateral temporomandibular joint (TMJ) arthroscopy

Received intraoperative platelet-rich plasma (PRP) or platelet-rich fibrin (PRF) injection during TMJ arthroscopy

Exclusion Criteria:

Age younger than 18 years or older than 75 years

Did not undergo TMJ arthroscopy

Did not receive intraoperative PRP or PRF injection

Incomplete clinical or follow-up data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 to 75 years who underwent unilateral or bilateral temporomandibular joint arthroscopy at a single institution. All patients received intraoperative intra-articular injection of platelet-rich plasma (PRP) or platelet-rich fibrin (PRF) as part of routine clinical care. This is a retrospective observational study based on review of existing medical records, with no prospective recruitment or intervention.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
pain intensity | from baseline to 6 months post-surgery.
  The primary endpoint of the study is the change in pain intensity from baseline to 6 months post-surgery.

SECONDARY OUTCOMES:
maximum unassisted opening (MMO) | baseline and various follow-up times in 6 months.
  collect data about maximum unassisted opening (MMO)

CONTACTS AND LOCATIONS:
Locations (1):
- Meikun Wang, Boston, Massachusetts, United States